CLINICAL TRIAL: NCT00859664
Title: Use of Pharmacogenetics in the Treatment of Children With Autistic Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Ilan Youngster, Assaf harofeh medical center
Other Study IDs: 145/07
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Autism; Neuroleptic Treatment
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Neuroleptics: Children with autistic spectrum disorder, treated with neuroleptics
  Interventions: Other: Genotyping of Cytochrome P450

INTERVENTIONS:
Other: Genotyping of Cytochrome P450 — Genotyping of Cytochrome P450

SUMMARY:
Children with autism are often treated with psychiatric drugs. These medications have been shown to improve their language and social function, and are important in improving their quality of life. In many cases it is difficult to determine the best drug dose, and a favorable response occurs in only 30%-70% of individuals, with many children suffering significant adverse drug reactions.

Pharmacogenetics is the study of the role of different genes on drug behavior. The cytochrome P450 is the most important enzyme, involved in the metabolism of a vast number of drugs, including psychiatric medications. The multiple variations in this gene can result in the different response observed in different patients, even when treated with similar doses of the drug.

Hypothesis(es):

Mapping the different types of cytochrome P450 gene, in children with autistic disorders will improve the rate of success of medical treatment, and prevent adverse drug reactions.

Potential Impact:

If successful, our study can help thousands of children and their families by developing a system of "tailored medicine" that is based on the specific activity of the various enzymes present in that particular patient. Better medical treatment will facilitate better daily interactions with the children and enhance their quality of life. Furthermore, recognizing children that are resistant to medication will prevent unnecessary use of drugs.

It should be noted this is the first study focusing on children receiving psychiatric medications using pharmacogenetics. Found to be effective, this method can also be applied to other groups of medications and to other patients.

ELIGIBILITY:
Inclusion Criteria:

* Age> 3 years
* Diagnosed with autism
* Treated with neuroleptics

Exclusion Criteria:

* Patients with known allergy to second generation neuroleptics.
* Patients with moderate to severe renal insufficiency
* Patients with liver disease
* Patients with active cardiac disease
* Patients with hypertension not responsive to anti-hypertensive therapy
* Patients with substance abuse
* Suicidal patients

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children over the age of 3, diagnosed with autism, treated with neuroleptics
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Genotyping of the polymorphic cytochrome P450 (CYP) 2D6 gene, in children with autistic spectrum disorder treated with neuroleptics, will improve treatment efficacy and prevent undesired adverse drug reactions. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical center, Ẕerifin, Israel